CLINICAL TRIAL: NCT00002888
Title: A RANDOMIZED PHASE III EVALUATION OF PACLITAXEL + G-CSF + CISPLATIN VERSUS CISPLATIN + 5-FU IN ADVANCED HEAD AND NECK CANCER
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065210; E-1395; SWOG-E1395
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2007-05

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether cisplatin plus fluorouracil are more effective than paclitaxel plus cisplatin in treating patients with advanced head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens in treating patients with advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the response rate, toxicity, quality-of-life, and overall survival at 1 year in patients with advanced head and neck carcinomas when treated with paclitaxel and cisplatin vs cisplatin and fluorouracil. II. Compare these regimens in terms of quality of life and correlate quality of life to toxicity in these patients. III. Compare these regimens in terms of pain intensity and correlate pain with quality of life and toxicity in these patients.

OUTLINE: This is a randomized study. Patients are stratified by disease status, performance status, and participating institution. Patients are randomized to one of two treatment arms. Arm I: Patients receive cisplatin IV over 30-120 minutes on day 1 and fluorouracil IV over 96 hours on days 1-4. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Arm II: Patients receive paclitaxel IV over 3 hours followed by cisplatin IV over 30-120 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Treatment continues until 2 courses past complete response (minimum of 6 courses). Patients with stable disease may discontinue treatment after 6 courses. Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 212 patients will be accrued for this study over 2.25 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous cell carcinoma of the head and neck considered incurable by surgery or radiotherapy Newly diagnosed extensive locoregional disease or distant metastases Locoregionally recurrent or persistent disease, or distant metastases occurring after initial surgery or radiotherapy No nasopharyngeal carcinoma No history of brain metastases Measurable or evaluable disease Documented progressive disease or biopsy-proven residual carcinoma required if sole measurable site previously irradiated

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Hematopoietic: ANC at least 1,500/mm3 Hemoglobin at least 10 g/dL (transfusion allowed) Hepatic: Bilirubin less than 1.5 mg/dL AST/ALT no greater than twice normal Alkaline phosphatase no greater than twice normal Renal: Creatinine no greater than 1.2 mg/dL OR Creatinine clearance at least 50 mL/min Calcium normal No history of hypercalcemia Cardiovascular: No congestive heart failure No serious arrhythmia requiring medication No myocardial infarction within 6 months No medications known to alter cardiac conduction (i.e., lanoxin, beta or calcium channel blockers) Other: No significant detectable or occult infection Complete evaluation required if elevated WBC (12,000 or greater) or fever (101.6 F or higher) No hypersensitivity to E. coli-derived proteins No allergy to drugs utilizing Cremophor No other malignancy within 3 years except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant Negative pregnancy test Fertile patients must use effective contraception Must complete quality of life and pain assessments at required intervals

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for recurrent disease At least 12 months since induction or neoadjuvant chemotherapy with paclitaxel or fluorouracil (6 months since cisplatin) Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Recovered from major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-03; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene A. Forastiere, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Maha Hadi A. Hussain, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (87):
- United States (87):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Ozarks Regional, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Hospital Tumor Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Gibson MK, Li Y, Murphy B, Hussain MH, DeConti RC, Ensley J, Forastiere AA; Eastern Cooperative Oncology Group. Randomized phase III evaluation of cisplatin plus fluorouracil versus cisplatin plus paclitaxel in advanced head and neck cancer (E1395): an intergroup trial of the Eastern Cooperative Oncology Group. J Clin Oncol. 2005 May 20;23(15):3562-7. doi: 10.1200/JCO.2005.01.057. PMID 15908667
- [Result] Argiris A, Li Y, Forastiere A, et al.: Prognostic factors and long-term survivorship in patients with recurrent or metastatic head and neck cancer (HNC): an analysis of two Eastern Cooperative Oncology Group (ECOG) randomized trials. [Abstract] J Clin Oncol 22 (Suppl 14): A-5514, 491s, 2004.
- [Result] Argiris A, Li Y, Forastiere A. Prognostic factors and long-term survivorship in patients with recurrent or metastatic carcinoma of the head and neck. Cancer. 2004 Nov 15;101(10):2222-9. doi: 10.1002/cncr.20640. PMID 15452834
- [Result] Wells N, Murphy B, Dietrich M, et al.: Quality of life and pain assessment for head and neck cancer patients treated on E1395: a comparison of two different cisplatin-based chemotherapy regimens. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-907, 2002.
- [Result] Murphy B, Li Y, Cella D, et al.: Phase III study comparing cisplatin (C) & 5-flourouracil (F) versus cisplatin & paclitaxel (T) in metastatic/recurrent head & neck cancer (MHNC). [Abstract] Proceedings of the American Society of Clinical Oncology 20; A-894, 2001.